CLINICAL TRIAL: NCT05455788
Title: Prosthetic Valve Sweing Ring Injection by Antiboitics Can Affect the Rate of Postoperative Infective Endocarditis?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Ibrahim Osman, Principle investigator, Assiut University
Other Study IDs: AssiutMedic
Record Dates: First submitted 2022-07-01; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Prosthetic Valve Endocarditis
MeSH Terms: interventions — Aminoglycosides

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing Cardiac valve replacement
  Interventions: Drug: Aminoglycoside

INTERVENTIONS:
Drug: Aminoglycoside — injection of sewing ring of prosthetic valve with aminoglycoside

SUMMARY:
Follow-up of patients undergoing cardiac valve replacements with prosthetic valve after injection of sewing ring of prosthetic valve with aminoglycoside for prevention of infective endocarditis.

ELIGIBILITY:
Inclusion Criteria:

* patients who need cardiac valve replacement for rheumatic or degenerative causes

Exclusion Criteria:

* Patients undergoing open heart surgery for any cause other than valve replacement
* patients who are younger than 20 years old.
* Patients undergoing valve repair.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with heart valve disease and indicated for valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
number of patients diagnosed with Infective endocarditis post valve replacement | 6 months post operative
  percentage of post operative clinical and echocardiographic diagnosis of infective endocarditis on prosthetic valve

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No